CLINICAL TRIAL: NCT01082094
Title: An Open Label Dose Escalation Study to Evaluate the Safety of a Single Escalating Dose of ACRX-100 Administered by Endomyocardial Injection to Cohorts of Adults With Ischemic Heart Failure
Brief Title: Study to Evaluate the Safety of a Single Escalating Dose of ACRX-100 in Adults With Ischemic Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Juventas Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JTCS-001
Record Dates: First submitted 2010-03-04; First posted 2010-03-08 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Heart Failure
Keywords: Ischemic heart failure; Congestive heart failure; Stromal cell-derived factor 1; SDF-1; Gene therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACRX-100 (Experimental): Cohort 1 = Low dose
  Cohort 2 = Middle dose
  Cohort 3 = High Dose
  Interventions: Biological: ACRX-100

INTERVENTIONS:
Biological: ACRX-100 — Three cohorts (16 total subjects) will be studied. There will be no concurrent controls. The dose will be escalated by increasing the total amount of ACRX-100 delivered per subject from low dose (n=4 subjects) to middle dose (n=6 subjects) to high dose (n=6 subjects). ACRX-100 will be injected directly into the myocardium as a single dose at multiple sites through a percutaneous, left ventricular approach using a needle injection catheter.

SUMMARY:
The purpose of this Phase 1 study is to assess the safety, tolerability, and preliminary efficacy of single escalating doses of ACRX-100 delivered via endomyocardial injection in adults with ischemic heart failure.

DETAILED DESCRIPTION:
This open label, 16 subject, Phase 1 dose-escalation study will demonstrate the initial safety of using ACRX-100 to treat heart failure in subjects with ischemic cardiomyopathy. Safety will be tracked at each dose by documenting all adverse events (AEs), with the primary safety endpoint being the number of major cardiac AEs at 30 days. In each cohort (n=4 in low dose, n=6 each in mid and high dose), subjects will receive a single dose of ACRX-100. Preliminary efficacy will be evaluated by measuring the impact on cardiac function via standard echocardiography measurements, cardiac perfusion via SPECT imaging, and improvement in NYHA classification.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* NYHA Class III
* Ischemic cardiomyopathy without an acute coronary syndrome within the last 6 months
* Residual well-demarcated region of LV systolic dysfunction defined as at least 3 consecutive segments of abnormal wall motion by echocardiography read at the echocardiography core laboratory
* LVEF less than or equal to 40% measured by echocardiography read at the echocardiography core laboratory
* No left ventricular wall thickness less than 0.5 cm measured by echocardiography read at the echocardiography core laboratory
* Mitral regurgitation of 0-2+ (inclusive) measured by echocardiography read at the echocardiography core laboratory
* Subject has an implanted, functional AICD
* Subject receiving stable optimal pharmacological therapy defined as:

  * ACE inhibitor and/or ARB, and Beta-blocker for 90 days with stable dose for 30 days unless contraindicate
  * Diuretic in subjects with evidence of fluid retention ASA unless contraindicated
  * Statin unless contraindicated
  * Aldosterone antagonist per physician discretion unless contraindicated
* Subjects with found diagnosis of diabetes must have had an ophthalmologist exam within the last year showing no active proliferative retinopathy

Exclusion Criteria:

* Planned revascularization within 30 days following enrollment
* Estimated Glomerular Filtration Rate < 30 ml/min*
* Inability to undergo SPECT imaging
* History of aortic valve regurgitation > 2
* Moderate/Severe aortic stenosis defined as AVA <1.5 cm2
* Presence of an artificial aortic valve
* Subjects with aortic aneurysm >3.8 cm
* History of cancer with exception of basal cell carcinoma and following results on age appropriate cancer screenings
* Subjects with persistent atrial fibrillation (per ACC/AHA/ESC guidelines, defined as recurrent AF episodes lasting longer than 7 days)
* Subjects with Biventricular pacing device implant within the last 3 months OR previously implanted Biventricular pacing device with programming planned to be reoptimized following enrollment in this trial
* Previous solid organ transplant
* Subjects with greater than 40% univentricular RV Pacing
* Subjects with uncontrolled diabetes defined as HbA1c >9.0%
* Participation in an experimental clinical trial within 30 days prior to enrollment
* Life expectancy of less than 1 year
* Positive pregnancy test (serum βHCG) in women of childbearing potential and/or unwillingness to use contraceptives or limit sexual activity
* Unwillingness of men capable of fathering a child to agree to use barrier contraception or limit sexual activity
* Subjects who are breast feeding
* Subjects with a positive test results for hepatitis B/C and/or HIV
* Total Serum Bilirubin >4.0 mg/dl
* Aspartate aminotransferase (AST) > 120 IU/L
* Alanine aminotransferase (ALT) > 135 IU/L
* Alkaline phosphatase (ALP): >300 IU/L
* Clinically significant elevations in PT or PTT relative to laboratory norms
* Proteinuria > 3.5 g/L
* Any subject with a known existing LV thrombus or has an LV thrombus detected during the screening period of this study. Presence of LV thrombus will be determined by echocardiography and the addition of echo-contrast if any question remains after non-contrast echocardiogram.
* History of drug or alcohol abuse within the last year
* A subject will be excluded if he/she is unfit for the trial based on the discretion of the site Principal Investigator

  * Estimated Glomerular Filtration Rate (eGFR) in ml/min is calculated using the subject's serum creatinine value with the following equation : eGFR = 186 x (serum creatinine in mg/dl)-1.154 x (Age)-.2303 x (Age) x (1.210 if subject is black) x (0.742 if subject is female)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of Major Adverse Cardiac Events (MACE) at 30 days post-injection | 30 days post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Losordo, MD, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Cardiology, PC, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Columbia University Medical Center, New York, New York